CLINICAL TRIAL: NCT02799199
Title: Fingolimod Real World Experience: the French Grand-Est Cohort
Acronym: Gilenya
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO14105
Record Dates: First submitted 2016-05-27; First posted 2016-06-14 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
Objectives: This study describes efficacy and safety of Fingolimod in patients treated for at least 6 months in the east of France from January 2011 to December 2014.

Background: The Grand-Est is a geographical region in France with a high prevalence of multiple sclerosis (more than 10000 patients registered in the European Database for Multiple Sclerosis (EDMUS) database). In this region and since January 2011, more than 1014 patients have been treated for at least 6 months with Fingolimod, the first oral therapy for patient with very active relapsing-remitting MS.

Methods: Features of patients followed up in the Grand-Est region and treated with fingolimod in the 6 university hospitals, general hospitals and private neurologists were reviewed in a retrospective study after identification of the clinical files reported in the EDMUS database.

ELIGIBILITY:
Inclusion Criteria:

* Patients with MS treated with Gilenya because of the disease

Exclusion Criteria:

* contraindications of Gilenya treatment or receiving Gilenya after the 31st of March 2014

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients treated with fingolimod for at least 6 months
Sampling Method: Probability Sample
Enrollment: 1014 (Actual)
Dates: Start 2014-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
the course of the disease by magnetic resonance imaging (MRI) | assessed between January 2012 and September 2014, up to a total of 32 months